CLINICAL TRIAL: NCT06704594
Title: Allopregnanolone and Dynamic GABA-A Receptor Plasticity in Selective Serotonin Reuptake Inhibitor Responsive Premenstrual Dysphoric Disorder
Acronym: BLOOM
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00445770; R01MH134904 (NIH)
Record Dates: First submitted 2024-11-21; First posted 2024-11-26 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Premenstrual Dysphoric Disorder (PMDD)
Keywords: pmdd; premenstrual dysphoric disorder; pms; premenstrual symptoms; premenstrual syndrome; blood draw; sertraline; ssri; mood symptoms; women; women with pms; women with pmdd; luteal phase; follicular phase; womens reproductive mental health; womens health; womens reproductive health; menstrual cycle; menses; periods; allopregnanolone; neuroactive steroids; inflammatory markers; epigenetics
MeSH Terms: conditions — Premenstrual Dysphoric Disorder; Premenstrual Syndrome | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants delegated to the "control" arm will be individuals without premenstrual symptoms in the luteal phase of the menstrual cycle. Participants will be asked to track mood across the menstrual cycle, answer self-report surveys, and complete four blood draws.
- PMDD with sertraline (Active Comparator): Participants delegated to the "PMDD with sertraline" arm will be individuals with severe premenstrual symptoms in the luteal phase of the menstrual cycle. Participants will be asked to track mood across two menstrual cycles, answer self-report surveys, and complete eight blood draws (four in each menstrual cycle). In the second cycle, participants in this arm will take a daily pill of 50 mg of sertraline from ovulation until menses onset (end of menstrual cycle 2).
  Interventions: Drug: sertraline 50 mg daily
- PMDD with placebo (Placebo Comparator): Participants delegated to the "PMDD with placebo" arm will be individuals with severe premenstrual symptoms in the luteal phase of the menstrual cycle. Participants will be asked to track mood across two menstrual cycles, answer self-report surveys, and complete eight blood draws (four in each menstrual cycle). In the second cycle, participants in this arm will take a daily placebo pill from ovulation until menses onset (end of menstrual cycle 2).
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: sertraline 50 mg daily — The intervention will be in the form of an oral pill, taken daily, from the day of positive urine ovulation test result until the day of menses onset.
  Arms: PMDD with sertraline
Drug: Placebo Oral Tablet — The placebo oral tablet will be of the same shape, color, and manufacturer as the sertraline 50 mg oral tablets. Tablet will be taken daily, from the day of positive urine ovulation test result until the day of menses onset.
  Arms: PMDD with placebo

SUMMARY:
Premenstrual dysphoric disorder (PMDD) is a severe affective disorder impacting millions of women worldwide, thought to be due to altered sensitivity to hormone fluctuations across the menstrual cycle. Neuroactive steroid hormones (NAS) and the gamma-aminobutyric acid (GABA)-A receptor (GABAAR) are thought to play a role in PMDD. This research will assess the blood levels of GABAergic NAS, expression of associated enzymes, and expression of GABAAR subunits across the premenstrual (luteal) phase of the menstrual cycle in healthy controls and individuals with PMDD. Within the PMDD group, the investigators will assess how these measures are affected by a low-dose antidepressant medication versus placebo. The results will provide a comprehensive view of the changes in these systems across the menstrual cycle and will add to the investigator's understanding of the mechanisms that underlie PMDD, as well as therapeutic mechanisms of PMDD treatment.

ELIGIBILITY:
Inclusion Criteria:

* female sex,
* fluent in the English language
* regular menstrual cycles (24-35 days)
* age 18-50 years old
* ability to give written informed consent

Exclusion Criteria:

* psychiatric medication use in the past 2 months
* substance use disorder in the past 6 months
* lifetime history of psychotic disorder including schizophrenia
* schizoaffective disorder, major depression with psychotic features
* history of psychiatric disorder other than PMDD in past year
* active suicidal ideation with plan or attempt in past 6 months
* steroid hormone or hormonal contraceptive use (except levonorgestrel as emergency contraceptive) in past 2 months
* pregnancy in past 6 months
* history of brain injury
* current or history of endocrine disorder including uncontrolled diabetes or thyroid disease
* BMI>40
* History of arrythmias, severe liver impairment, history of seizure disorder
* If currently taking the following meds: methylene blue, linezolid
* Other prohibited concomitant meds are Monoamine oxidase inhibitors (MAOIs), pimozide, and disulfiram

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 288 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Neuroactive Steroid Levels | Post ovulation up to 2 days, up to 5 days pre-menses prediction
  The primary outcome variable is levels of neuroactive steroids in blood; from the early luteal phase (2 days post ovulation) compared to the late luteal phase (days 5 to 1 prior to predicted menses onset)

SECONDARY OUTCOMES:
Neurosteroidogenic enzyme expression levels | First menstrual cycle, up to 3 months
  Neurosteroidogenic enzyme expression levels will be measured in the early luteal phase (2 days post ovulation) and the late luteal phase (days 5 to 1 prior to predicted menses onset). Levels will be compared between the healthy controls and PMDD groups at cycle 1, and between sertraline and placebo groups at cycle 2, respectively; between cycle 1 (first menstrual cycle when blood draws will be completed) and until the end of the participants' time on the study (2-3 months).
GABAAR subunit expression levels | first menstrual cycle, up to 3 months
  GABAAR subunit expression will be measured in the early luteal phase (2 days post ovulation) and the late luteal phase (days 5 to 1 prior to predicted menses onset). The investigators will compare GABAAR subunit expression levels between controls and PMDD groups at L1, and between sertraline and placebo groups at L2, respectively; between cycle 1 (first menstrual cycle when blood draws will be completed) and until the end of the participants' time on the study (2-3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Liisa Hantsoo, PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Reproductive Mental Health Center, Baltimore, Maryland
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No